CLINICAL TRIAL: NCT07354178
Title: Randomized Clinical Trial to Assess Hemostasis by Applying Collagen-based Thrombin-containing Hemostat in Spinal Surgery
Brief Title: Study of Collagen-Based Thrombin Hemostat for the Control of Bleeding in Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DALIM TISSEN Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRT-CS01
Record Dates: First submitted 2025-11-24; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Spinal Tumor; Spinal Injury; Hemostasis; Spinal Stenosis; Spinal Surgery; Intraoperative Bleeding
MeSH Terms: conditions — Spinal Cord Neoplasms; Spinal Injuries; Spinal Stenosis; Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Group applied with CollaStat®
  Interventions: Device: Floseal®
- Control Group (Active Comparator): Group applied with Floseal®
  Interventions: Device: CollaStat®

INTERVENTIONS:
Device: CollaStat® — Clinical subjects are enrolled after the clinical investigator confirms that there are bleeding sites where hemostasis by normal procedures (compression, suturing, electrosurgical scalpel, etc.) is ineffective or difficult to perform. To arrest intraoperative bleeding, the study group is treated with Dalim Tissen's CollaStat® and compressed with general gauze.
  Arms: Control Group
Device: Floseal® — Clinical subjects are enrolled after the clinical investigator confirms that there are bleeding sites where hemostasis by normal procedures (compression, suturing, electrosurgical scalpel, etc.) is ineffective or difficult to perform. To arrest intraoperative bleeding, the control group is treated with Baxter's Floseal® and compressed with general gauze
  Arms: Study Group

SUMMARY:
This clinical trial evaluates the effectiveness and safety of a collagen-based hemostatic agent containing thrombin in patients undergoing spinal surgery. The study compares this investigational product with an existing hemostatic agent to assess whether it performs equally well in controlling surgical bleeding. Patients with spinal stenosis, tumors, or trauma who require spinal surgery will be enrolled. The hemostat will be applied intraoperatively when grade 3 bleeding is observed. The study aims to determine how well the product works in achieving hemostasis and its safety when it is used during surgery.

DETAILED DESCRIPTION:
This was a randomized, single-blind, active-controlled clinical trial designed to assess the non-inferiority of a collagen-based thrombin-containing topical hemostat (CollaStat) compared to an existing hemostatic agent (Floseal) in patients undergoing spinal surgery. The investigational product was designed to be highly biocompatible to reduce adverse effects in case of in-body residue after application. Patients who underwent spinal surgery due to spinal stenosis, tumors, or trauma were enrolled and randomized in a 1:1 ratio. The hemostatic products were applied intraoperatively at bleeding sites classified as grade 3. For grade 4 or 5 bleeding, temporary hemostatic procedures were performed first to reduce bleeding intensity before applying the assigned hemostat. The study's primary endpoint was the hemostasis success rate, defined as the achievement of hemostasis within 1 minute, 2 minutes, 3 minutes, 6 minutes, and 10 minutes of product application without additional intervention. Secondary outcomes included time to hemostasis, number of hemostatic units used per patient, volume of postoperative surgical drainage, length of hospital stay, incidence of intraoperative rebleeding, occurrence of postoperative hematoma or surgical site infection, and overall hemostatic effect assessed across all treated bleeding sites.

ELIGIBILITY:
Inclusion Criteria:

1. An individual who has voluntarily signed the written consent form for participating in the research as a trial subject
2. Patients aged 20 or older
3. Patients who are able to participate throughout the entire clinical trial period
4. Patient scheduled to have spinal surgery due to spinal stenosis, spinal tumor, injury, etc.
5. Patients for whom hemostasis is difficult to achieve using standard procedures
6. Patients with grade 3 or higher bleeding * Grade 4 or 5 bleeding is reduced to grade 3 by normal procedures (compression, sutures, electrosurgical scalpel, etc.).

Exclusion Criteria:

1. Pregnant women or those planning to become pregnant within 1 month after application of the collagen-based hemostat
2. Individuals with hypersensitivity to bovine-, porcine-, or animal-derived materials
3. Individuals deemed inappropriate for participation by the investigators
4. Patients who are using treatments that may affect the test results
5. Patients with active infections at the surgical site
6. Patients with contraindications to the use of local hemostatic materials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Hemostasis success rate | Hemostasis at the first bleeding site is confirmed at 1 minute, 2 minutes, 3 minutes, 6 minutes, and 10 minutes
  After applying the haemostatic agent to the bleeding site, gentle compression is performed using surgical gauze. After lifting the gauze and washing off the excess hemostatic agent, check if hemostasis is maintained

SECONDARY OUTCOMES:
Time to hemostasis | Intraoperation
  Record the time point when hemostasis is achieved.
Number of hemostats used | Intraoperation
  Record the number of hemostats used until hemostasis.
Length of Hospital Stay | From the date of surgical operation (Visit 2) until the date of hospital discharge, assessed up to 1 week (±3 days) after surgery
  Length of hospital stay is defined as the number of days from the date of surgery (Visit 2) to the date of hospital discharge.
Incidence of adverse events | From first application of the investigational medical device through end of follow-up (up to 8 weeks post-surgery)
  Adverse events include hematoma and infection.
Drain amount | 3 days after surgery
  Record the drain amount until the 3rd postoperative day.
Presence of rebleeding at the index bleeding site | From first application (Visit 2; day of surgery) through end of follow-up (up to 8 weeks post-surgery)
Evaluation of Handling Characteristics (as Assessed by the Surgeon) | Intraoperative
  Hemostasis will be assessed intraoperatively at all treated bleeding sites after application of the investigational product (IP). Only the assigned IP should be used for the same patient.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Yongin Severance Hospital, Yongin-si, Giheung-gu
  - Severance Hospital, Yonsei University Health Syetem, Seoul, Seodaemun-gu

IPD SHARING:
Plan to Share IPD: Undecided
Undecided. The plan for sharing individual participant data has not yet been determined.